CLINICAL TRIAL: NCT04819789
Title: Digestibility of Fermotein™
Acronym: MyDi
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wageningen University and Research (Other)
Collaborators: The Protein Brewery (Unknown)
Responsible Party: Principal Investigator, Diederik Esser, Project leader clinical trials, Wageningen University and Research
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Other
Other Study IDs: NL74595.081.20
Record Dates: First submitted 2021-03-24; First posted 2021-03-29 (Actual); Last update posted 2021-05-25 (Actual); Status verified 2021-05

CONDITIONS: Digestive System
Keywords: Fermotein™; Digestibility; Protein digestion kinetics; Mycoprotein

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Fermotein™ dry (Experimental): Fermotein™ powder presented in the form of a porridge.
  Interventions: Other: Fermotein™ dry powder porridge
- Fermotein™ wet (Experimental): Fermotein™ wet presented in the form of a porridge.
  Interventions: Other: Fermotein™ wet porridge
- Fermotein™ modified wet (Experimental): Fermotein™ modified wet presented in the form of a porridge.
  Interventions: Other: Fermotein™ modified wet porridge
- Mycoprotein (Active Comparator): This mycoprotein product presented in the form of a porridge.
  Interventions: Other: Mycoprotein porridge (matching control)

INTERVENTIONS:
Other: Fermotein™ dry powder porridge — At one out of four test days: Fermotein™ dry powder mixed with water and a few drops of food grade flavor concentrates, to obtain a porridge representing a 20g protein load.
  Arms: Fermotein™ dry
Other: Fermotein™ wet porridge — At one out of four test days: Fermotein™ wet mixed with water and a few drops of food grade flavor concentrates, to obtain a porridge representing a 20g protein load.
  Arms: Fermotein™ wet
Other: Fermotein™ modified wet porridge — At one out of four test days: Fermotein™ modified wet mixed with water and a few drops of food grade flavor concentrates, to obtain a porridge representing a 20g protein load.
  Arms: Fermotein™ modified wet
Other: Mycoprotein porridge (matching control) — At one out of four test days: Mycoprotein (Quorn) mixed with water and a few drops of food grade flavor concentrates, to obtain a porridge representing a 20g protein load.
  Other Names: Quorn
  Arms: Mycoprotein

SUMMARY:
This study aims to assess the degree of digestibility of 3 different Fermotein™ products and compare this to a reference commercially available Mycoprotein (Quorn) and to assess the effects on blood glucose and insulin levels.

The study has a randomized, cross-over, double blind, controlled design. Four different treatments, all representing a 20g protein load, will be evaluated with a washout period of minimum one week between the test days. On test days, research subjects will receive a product e.g. Fermotein™ dry, Fermotein™ wet, modified Fermotein™ wet and a reference Mycoprotein (Quorn), in the form of a porridge, in randomized order. Blood will be collected via a catheter before and up-to five hours after protein consumption. Wellbeing, health complaints or other adverse effects will be collected via short questionnaires during each test day. After each test day gastrointestinal complaints are collected via an online questionnaire.

DETAILED DESCRIPTION:
Mycoprotein is a protein source derived from fungi produced for human consumption. It is high in protein, high in fiber, low in saturated fat and contains no cholesterol. Their functional properties and nutrient content make them ideal to use as an ingredient for meat alternatives. Fermotein™ is such a mycoprotein type novel food source. The digestion characteristics of Fermotein™ are not known, but essential to evaluate their future potential as a sustainable protein source. Also, information on the degree of digestibility would strengthen a novel food dossier that is being constructed for this product.

The primary objective is to assess the degree of digestibility of 3 different Fermotein™ products and compare this to a reference commercially available Mycoprotein (Quorn). Secondary objectives are to assess the effects on blood glucose and insulin levels.

The study has a randomized, cross-over, double blind, controlled design. Four different treatments, all representing a 20g protein load, will be evaluated with a washout period of minimum one week between the test days. On test days, research subjects will receive a product e.g. Fermotein™ dry, Fermotein™ wet, modified Fermotein™ wet and a reference Mycoprotein (Quorn), in the form of a porridge, in randomized order. Blood will be collected via a catheter before and up-to five hours after protein consumption. Wellbeing, health complaints or other adverse effects will be collected via short questionnaires during each test day. After each test day gastrointestinal complaints are collected via an online questionnaire.

ELIGIBILITY:
Inclusion Criteria:

* Apparently healthy men and women;
* Age between 18 and 70 years;
* Body mass index (BMI) between 18.5 and 30 kg/m2 ;
* Having veins suitable for blood sampling via a catheter (judged by study nurse/ medical doctor).

Exclusion Criteria:

* Any metabolic, gastrointestinal, inflammatory or chronic disease (such as diabetes, anaemia, hepatitis, cardiovascular disease),or having a condition or disease that may lead to an impaired immune system
* History of gastrointestinal surgery or having (serious) gastrointestinal complaints;
* History of liver dysfunction (cirrhosis, hepatitis) or liver surgery;
* Kidney dysfunction (self-reported);
* Any use of medication that may suppress the immune system, this will be judged by the medical supervisor;
* Use of medication that may influence the study results, such as gastric acid inhibitors, laxatives, stomach protectors and drugs that can affect intestinal motility, this will be judged by the medical supervisor;
* Anaemia (Hb values <7.5 mmol/L for women and <8.5 mmol/L for men);
* Reported slimming, medically prescribed or other extreme diets;
* Not willing to give up blood donation during the study;
* Current smokers;
* Alcohol intake ≥4 glasses of alcoholic beverages per day;
* Pregnant, lactating or wishing to become pregnant in the period of the study (self-reported);
* Abuse of hard drugs;
* Having food allergies;
* Not having a general practitioner;
* Participation in another clinical trial at the same time;
* Being an employee of the department Food, Health & Consumer Research of Wageningen Food & Biobased Research.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2021-04-13 (Actual); Primary Completion 2021-05-20 (Actual); Study Completion 2021-05-20 (Actual)

PRIMARY OUTCOMES:
Change in degree of digestibility | During the intervention period on 4 test days: at baseline and postprandial blood samples will be collected from the cannula at 10 time points (T=0, 30, 60, 75, 90, 120, 150, 180, 240, 300 minutes).
  In order to assess change in the degree of digestibility, we determine 19 free amino acids in blood samples collected via a catheter before and at several time points up-to five hours after protein source consumption. Blood amino acids will be determined by the laboratory of Wageningen FBR, according a valid method: AccQ-Tag ultra-derivation kit & HPLC.

SECONDARY OUTCOMES:
Change in plasma glucose levels | During the intervention period on 4 test days: at baseline and postprandial blood samples will be collected from the cannula at 9 time points (T=0, 30, 60, 90, 120, 150, 180, 240, 300 minutes).
  Plasma glucose levels will be determined in blood samples collected via a catheter before and at several time points up-to five hours after protein source consumption (hospital laboratory Ziekenhuis Gelderse vallei, Ede, the Netherlands).
Change in plasma insulin levels | During the intervention period on 4 test days: at baseline and postprandial blood samples will be collected from the cannula at 9 time points (T=0, 30, 60, 90, 120, 150, 180, 240, 300 minutes).
  Plasma insulin levels will be determined in blood samples collected via a catheter before and at several time points up-to five hours after protein source consumption (hospital laboratory Ziekenhuis Gelderse vallei, Ede, the Netherlands).

CONTACTS AND LOCATIONS:
Overall Officials: Diederik Esser, PhD, Principal Investigator — Wageningen University and Research
Locations (1):
- Stichting Wageningen Research, Wageningen, Gelderland, Netherlands

IPD SHARING:
Plan to Share IPD: No